CLINICAL TRIAL: NCT01087580
Title: A Randomized Phase-II Pilot Trial of Docetaxel and Prednisone Versus Radiation Therapy Plus Docetaxel and Prednisone in Patients With Nonmetastatic and Oligometastatic Castrate Resistant Prostate Cancer
Brief Title: Docetaxel + Prednisone With or Without Radiation for Castrate Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 08U3; STU0022442 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-03-03; First posted 2010-03-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: PROSTATE CANCER
Keywords: Prostate Cancer; non metastatic prostate cancer; oligometastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy alone, no radiation therapy (Experimental): A) Docetaxel: 75 mg/m2 IV infusion over 1 hour on day 1 of each cycle every 21 days
  B) Prednisone: 10 mg orally for 21 days after each dose of docetaxel
  Interventions: Drug: Docetaxel and Prednisone
- Chemotherapy with Radiation Therapy (Experimental): A) Docetaxel: 75 mg/m2 IV infusion over 1 hour on day 1 of each cycle every 21 days B) Prednisone: 10 mg orally for 21 days after each dose of docetaxel
  GROUPS 1 and 2 Whole Pelvis (45 Gy) + Prostate boost (20-25 Gy) in 1.8 Gy fractions, 5 fractions/week.
  GROUPS 2 Bone metastasis (bone scan index < 1.4%): 30 Gy in 10 fractions or 35 Gy in 12 fractions.
  GROUPS 1,2 Abdominal Nodes (IF POSITIVE ON CT/MRI SCAN): 45-50 Gy in 1.8 Gy fractions, 5 fractions/week.
  Interventions: Drug: Docetaxel and Prednisone; Drug: Radiation Therapy

INTERVENTIONS:
Drug: Docetaxel and Prednisone — A) Docetaxel: 75 mg/m2 IV infusion over 1 hour on day 1 of each cycle every 21 days B) Prednisone: 10 mg orally for 21 days after each dose of docetaxel
  Other Names: Taxotere
  Arms: Chemotherapy alone, no radiation therapy
Drug: Docetaxel and Prednisone — A) Docetaxel: 75 mg/m2 IV infusion over 1 hour on day 1 of each cycle every 21 days B) Prednisone: 10 mg orally for 21 days after each dose of docetaxel
  Other Names: Taxotere
  Arms: Chemotherapy with Radiation Therapy
Drug: Radiation Therapy — GROUPS 1 and 2 Whole Pelvis (45 Gy) + Prostate boost (20-25 Gy) in 1.8 Gy fractions, 5 fractions/week.
  GROUPS 2 Bone metastasis (bone scan index < 1.4%): 30 Gy in 10 fractions or 35 Gy in 12 fractions.
  GROUPS 1,2 Abdominal Nodes (IF POSITIVE ON CT/MRI SCAN): 45-50 Gy in 1.8 Gy fractions, 5 fractions/week.
  Arms: Chemotherapy with Radiation Therapy

SUMMARY:
The main purpose of this study is to find out whether adding radiation therapy to the standard treatment of chemotherapy for prostate cancer is tolerated well and is more effective than the standard treatment of chemotherapy alone

DETAILED DESCRIPTION:
Most physicians would consider chemotherapy to be the standard for prostate cancer. In this study all participants will receive the standard chemotherapy. In addition, half the participants will also receive radiation therapy. It is hoped that the radiation therapy will provide additional benefit. The use of radiation therapy and chemotherapy for patients with this kind of cancer is not considered standard treatment at the present time.

Participants will be randomized into groups (or Arms) by a computer program. Participants randomized to Arm 1 will receive chemotherapy alone. Participants in Arm 2 will receive chemotherapy and radiation therapy. Participants in both groups (Arm 1 and Arm 2) will receive standard chemotherapy with docetaxel and prednisone. Docetaxel is given through a needle in a vein in the arm every 3 weeks or 21 days. Participants will take a prednisone tablet once per day until 21 days after the last dose of docetaxel. In addition, all participants will be given a drug called dexamethasone twice daily for 6 doses to help with the side effects of docetaxel. Participants in Arm 2 will first receive radiation therapy to the pelvis and prostate gland. Radiation therapy will be delivered once a day, five days a week for a total of 8-9 weeks. Then beginning 4-6 weeks after the end of radiation therapy, chemotherapy will be given, as described above. In both Arms, the total number of cycles of docetaxel and prednisone will depend upon how the tumor responds to these drugs. All patients should receive a minimum of three cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of castrate resistant prostate cancer.
* Participants must be 18 years old or older.
* Biopsy of tissue from the prostate or enlarged lymph nodes may be required.
* Patients must sign study specific informed consent prior to study entry.
* Men of child-producing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months afterwards.

Exclusion Criteria:

* Participants cannot have prior chemotherapy for prostate cancer.
* Participants cannot have prior radiation therapy to the pelvis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Estimation of progression free survival(PFS) and response rate | Day one of each treatment cycle. cycles are every 21 days and at the end of post-treatment
  The primary objective is to estimate the progression free survival (PFS) and treatment response of patients with non-metastatic or oligometastatic CRPC in the two study arms of either chemotherapy alone (ARM 1) or a combination of RT and chemotherapy (ARM 2).

SECONDARY OUTCOMES:
Overall survival of patients | at study completion and during follow-up (At least every 3 months (12 weeks) until evidence of progression or relapse for a maximum of 2 years, subsequently every 4 months for 2 years, then every 6 months for 2 years from the time of registration)
  One secondary objective is to estimate the overall survival of patients with non-metastatic or oligometastatic castrate resistant prostate cancer in the two study arms of either chemotherapy alone (ARM 1) or a combination of RT and chemotherapy (ARM 2).
Multiple gene profiles will be analyzed. | At Study Completion
  Gene profiles using microarray techniques will be compared in order to identify genes important in governing the response to chemotherapy and radiation therapy in non-metastatic or oligometastatic castrate resistant prostate cancer. The expression and mutation of p53 gene, expression of androgen receptor (AR), PSA and neuroendocrine differentiation in non-metastatic or oligometastatic CRPC using immunohistochemical analysis will also be studied.
Measure of prostate antigen-specific immune response | Every 21 days during treatment. Follow-up is every 3 mo until evidence of progression or relapse for 2 years, then every 4 mo for 2 years, then every 6 mo for 2 years from the time of registration)
  This secondary objective will determine if treatment of patients with non-metastatic or oligometastatic castrate resistant prostate therapy with chemotherapy, with or without radiation therapy, elicits prostate antigen-specific immune responses.
Estimation of treatment-related toxicity | Every 21 days. weekly radiation therapy, Follow-up is every 3 mo until evidence of progression or relapse for 2 years, then every 4 mo for 2 years, then every 6 mo for 2 years from the time of registration
  This secondary objective will estimate the treatment-related toxicity of patients with non-metastatic or oligometastatic castrate resistant prostate cancer in the two study arms of either chemotherapy alone (ARM 1) or a combination of RT and chemotherapy (ARM 2).

CONTACTS AND LOCATIONS:
Overall Officials: John Kalapurakal, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Hematology Oncology Associates, Chicago, Illinois
  - Northwestern University, Northwestern Memorial Faculty Foundation, Chicago, Illinois